CLINICAL TRIAL: NCT07020598
Title: Effect of a Sepsis Alert Routine in the Emergency Department: A Before-and-After Cohort Study
Brief Title: Sepsis Alert Routine Implementation in the Emergency Department
Acronym: SARIED
Status: Completed | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristoffer Strålin, Associate Professor, Senior Consultant, Region Stockholm
Other Study IDs: 2017/1358-31; K 2017-2778 (Other: REGX_SE_REGION STHLM KAROLINSKA)
Record Dates: First submitted 2025-05-30; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Sepsis
Keywords: Sepsis; Emergency Department; Sepsis Alert; Antibiotics; Clinical Implementation; Mortality; Propensity Score Matching; Time to Treatment
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the impact of a structured sepsis alert routine, that has been implemented in the Emergency Department (ED) of Karolinska University Hospital Huddinge, Sweden. Using a retrospective cohort design, it compares patient outcomes before and after implementation of the routine. The main aim is to assess whether the sepsis alert system improves 28-day mortality among patients with suspected sepsis.

DETAILED DESCRIPTION:
Sepsis is a life-threatening condition associated with high morbidity and mortality, affecting millions of people globally each year. Timely recognition and early initiation of treatment are critical for improving outcomes. In response to this need, a structured sepsis alert routine was introduced in October 2017 at the Emergency Department (ED) of Karolinska University Hospital Huddinge, a large tertiary care hospital in Stockholm, Sweden.

The sepsis alert routine was designed to identify patients at risk of sepsis early in their ED visit, using predefined triage criteria. The alert was triggered by ED nurses based on suspected infection and specific triage parameters using the RETTS system (Rapid Emergency Triage and Treatment System). Patients with triage priority 1, or triage priority 2-3 combined with a blood lactate level of >3.2 mmol/L, were eligible. Once activated, a multidisciplinary response team-including physicians from the ED, Infectious Diseases, and Intensive Care Unit-was rapidly assembled to coordinate patient assessment and initiate early, protocolized sepsis care, including prompt antibiotic treatment and fluid resuscitation. The response followed a standardized checklist aligned with the Surviving Sepsis Campaign guidelines.

This study evaluates the clinical impact of the sepsis alert routine by comparing outcomes before and after its implementation. It uses a retrospective, observational cohort design with two data collection periods: a 2-year control period before the intervention (October 2015 - September 2017) and a 2.25-year period during which the sepsis alert was active (October 2017 - December 2019). All patients included were ≥18 years of age, admitted to hospital from the ED with suspected bacterial infection (defined by antibiotic therapy initiated within 48 hours and continued for at least 96 hours or until death, discharge, or ICU transfer), and met sepsis alert criteria.

To assess the effectiveness of the intervention, the primary outcome is 28-day all-cause mortality. Secondary outcomes include 90-day mortality, time to antibiotic administration, and length of hospital stay. Multivariable logistic regression will be used to analyze the full study population, with the intervention period (pre vs. post-implementation) as the main exposure variable, adjusting for covariates including sex, age, comorbidities (Charlson Comorbidity Index), SOFA score, triage priority, infection focus, body temperature, and do-not-resuscitate orders.

To further reduce confounding by indication, a propensity score matching analysis will be performed comparing patients who triggered the sepsis alert with matched historical controls. Propensity scores will be estimated using a logistic regression model including the aforementioned covariates as well as bacteremia status. Balance diagnostics and sensitivity analyses will be conducted to evaluate and account for any residual imbalances. Time-to-event outcomes will be analyzed using Kaplan-Meier survival curves.

This study will contribute important real-world data on the implementation of a sepsis alert system in a high-volume academic ED setting, and its potential to improve sepsis care and reduce mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Admitted to hospital via the Emergency Department
* Fulfillment of sepsis alert triage criteria (per RETTS system)
* Antibiotic therapy initiated within 48 hours and continued ≥96 hours or until death/discharge/ICU transfer, as marker for suspected bacterial infection

Exclusion Criteria:

* Readmission within 28 days of a previous eligible admission
* No antimicrobial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presented at the Emergency Department with triage criteria for sepsis alert and antibiotic therapy initiated within 48 hours and continued for at least 96 hours or until death, discharge, ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 3389 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28 days after presentation
  Death from any reason between presentation (day 0) to day 28

SECONDARY OUTCOMES:
90-day all-cause mortality | 90 days after presentation
  Death from any reason between presentation (day 0) and day 90
Lenght of hospital stay | From admission to discharge (up to 90 days after admission)
  Duration from admission to discharge
Time to first dose of antibiotics | From arrival to antibiotic administration (up to 48 hours from arrival)
  Time from arrival in the Emergency Department to antibiotic administration